CLINICAL TRIAL: NCT01585506
Title: Psychosocial Factors Related to Compliance With Treatment With Biphasic Insulin Analogues
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-4018
Record Dates: First submitted 2012-03-26; First posted 2012-04-26 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire responders
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Patients to complete the "WHO-5 Well-being Index" questionnaire
Other: No treatment given — Physicians to complete two questionnaires, "Demographic Data and Disease and Treatment Course" and "Questionnaire of Potential Difficulties in the Period of Treatment Switching from Insulin to Its Analogues"

SUMMARY:
This study is conducted in Europe. The aim of this study is to investigate psychosocial factors related to compliance with treatment with biphasic insulin analogues.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes in whom therapy with biphasic insulin analogues was started

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians who switched therapy from biphasic human insulins to a biphasic insulin analogue providing questionnaires for completion to patients whose therapy was switched from biphasic human insulins to biphasic insulin analogues
Sampling Method: Non-Probability Sample
Enrollment: 3618 (Actual)
Dates: Start 2010-09-20 (Actual); Primary Completion 2010-12-20 (Actual); Study Completion 2010-12-20 (Actual)

PRIMARY OUTCOMES:
Frequency and level of difficulty in introducing changes in compliance with the guidelines for biphasic insulin analogue use in subjects previously treated with biphasic human insulins | Up to 3 months

SECONDARY OUTCOMES:
Correlations between the difficulty in introducing changes in compliance with the guidelines for biphasic insulin analogue use in subjects previously treated with biphasic human insulins, and psychosocial factors | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Warsaw, Poland

REFERENCES:
- [Result] Kokoszka A. Treatment adherence in patients with type 2 diabetes mellitus correlates with different coping styles, low perception of self-influence on disease, and depressive symptoms. Patient Prefer Adherence. 2017 Mar 17;11:587-595. doi: 10.2147/PPA.S124605. eCollection 2017. PMID 28360512
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com